CLINICAL TRIAL: NCT04267055
Title: DISSECT-N (Dissection Navion Registry)
Brief Title: DISSECT-N Post Market Data Collection Registry
Acronym: DISSECT-N
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: NAMSA (Other)
Responsible Party: Sponsor
Other Study IDs: MDT19030 DISSECT-N
Record Dates: First submitted 2020-01-29; First posted 2020-02-12 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Aortic Dissection
MeSH Terms: conditions — Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Valiant Navion Thoracic Stent Graft System — Placement of the Valiant Navion for endovascular repair of a dissection in the thoracic aorta.

SUMMARY:
DISSECT-N is a post-market registry designed to assess real-world safety and effectiveness of Valiant Navion Thoracic Stent Graft System in the treatment of thoracic aortic dissections in real world practice.

DETAILED DESCRIPTION:
DISSECT-N is a prospective, observational, global, multi-center, post-market registry designed to assess real-world safety and effectiveness of Valiant Navion Thoracic Stent Graft System in the treatment of thoracic aortic dissections in real world practice.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years old
* Subject was treated in the last 7 days, or is intended to be treated, with the Valiant Navion Thoracic Stent Graft System for a dissection in the thoracic aorta
* Subject is willing to comply with standard of care clinical follow-up
* Subject or legal representative or consultee, as applicable has consented for study participation and signed the approved Informed Consent

Exclusion Criteria:

* Subject is participating in an investigational drug or device study which may bias or interfere with the endpoints and follow-up of this study.
* Subject is pregnant (not an exclusion if allowed per local regulatory requirements, pregnancy test to be performed where required)
* Subject has an active COVID-19 infection or relevant history of COVID-19. Relevant history of COVID-19 is defined as availability of a positive COVID-19 test with sequela or hospitalization for treatment of COVID-19. Subjects with a positive COVID-19 test who were asymptomatic or had mild symptoms should be excluded only if the positive test was less than 3 months prior to enrollment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population shall include all subjects diagnosed with a dissection of the thoracic aorta who have been treated, or are intended to be treated, with the Valiant Navion.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Composite safety and effectiveness | 1-month post index procedure
  Safety: Major Adverse Events (MAEs) Defined as: all-cause mortality (ACM), retrograde type A dissection (RTAD), aortic rupture, permanent paraplegia and paraparesis, stent induced new entry tear, conversion to open repair, disabling stroke, and non-preexisting renal failure.
  Effectiveness: Technical success defined as ability to advance, deploy and position the Valiant Navion Thoracic Stent Graft at target site with successful coverage and sealing of the proximal entry tear and removal of the delivery system.
  The primary endpoint is a dichotomous study outcome and a composite endpoint. A subject who has technical success and no MAE reported within 1-month will be considered a success.

SECONDARY OUTCOMES:
Aortic remodeling | 1-month, 1, 2 and 3 years
  Rate of aortic remodeling based on follow-up imaging.
Access related complications | peri-operative
  Rate of access related complications as proportion of evaluable patients.
Stent induced entry tear | 1, 2 and 3 years
  Rate of stent induced entry tear as proportion of evaluable patients.
Stent graft migration | 1, 2 and 3 years
  Rate of stent graft migration (>10mm) as proportion of evaluable patients.
Stent graft integrity | 1-month, 1, 2 and 3 years
  Rate of each type of loss of stent graft integrity (kink, twist, fracture, occlusion, or stenosis) as a proportion of evaluable patients based on follow-up imaging.
Disease progression | 1,2 and 3 years
  Extension of dissection.
Transient Ischemic Attack (TIA)/minor strokes | 1-month
  Rate of TIA/minor stroke as a proportion of evaluable patients.
Transient spinal cord ischemia | 1-month, 1, 2 and 3 years
  Rate of transient spinal cord ischemia as a proportion of evaluable patients.
Unplanned secondary procedures | 1, 2 and 3 years
  Rate of unplanned secondary procedures.
False lumen perfusion | 1-month, 1, 2 and 3 years
  Rate of each type of false lumen perfusion based on follow-up imaging.
Endoleaks | 1-month, 1, 2 and 3 years
  Rate of each type of endoleak based on follow-up imaging.
Major adverse events | 1, 2 and 3 years
  Major adverse events defined as:
  * All-cause mortality (ACM)
  * Retrograde type A dissection (RTAD)
  * Aortic rupture
  * Permanent paraplegia and paraparesis
  * Stent induced new entry tear
  * Conversation to open repair
  * Disabling stroke
  * Non-preexisting renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Ross Milner, MD, Principal Investigator — The University of Chicago Medicine & Biological Sciences
Locations (22):
- United States (12):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Michigan Health System - University Hospital, Ann Arbor, Michigan
  - Albany Medical Center, Albany, New York
  - Northwell Health Lenox Hill Hospital, New York, New York
  - Atrium Health's Carolinas Medical Center, Charlotte, North Carolina
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor Plano, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Rigshospitalet, Copenhagen, Denmark
- General Hospital of Athens, Evaggelismos, Athens, Greece
- Ospedale San Raffaele - Milano, Milan, Italy
- Japan (2):
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Keio University Hospital, Tokyo
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Auckland City Hospital, Grafton, New Zealand
- Narodny Ustav Srdcovych a Cievnych Chorob, A.S., Bratislava, Slovakia
- Severance Hospital, Seoul, South Korea
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No